CLINICAL TRIAL: NCT01296815
Title: Intralesional Bevacizumab for Treating AIDS-associated Kaposi´s Sarcoma of the Larynx, Pharynx and Oral Cavity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro de Investigación en. Enfermedades Infecciosas, Mexico (Other Government)
Responsible Party: Principal Investigator, Gustavo Reyes-Teran, Gustavo Reyes-Teran, Centro de Investigación en. Enfermedades Infecciosas, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C41-10
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Kaposi´s Sarcoma
Keywords: Kaposi sarcoma; HIV; Bevacizumab
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HAART (No Intervention): Patients received antiretroviral treatment according to the Guidelines for the Use of Antiretroviral Agents in HIV-1-Infected Adults and Adolescents
- HAART+ Bevacizumab injection (Experimental): Patients received antiretroviral treatment according to the Guidelines for the Use of Antiretroviral Agents in HIV-1-Infected Adults and Adolescents. Patients received 3 intralesional injections of bevacizumab (Avastin, Genentech, San Francisco, California) in the target lesion every 2 weeks. Bevacizumab was injected using an insulin syringe in a submucosal plane. The volume injected was based on the size of the target lesion; the dose was 0.2 mL (5 mg) per cm2.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Intralesional bevacizumab, dosis of 5mg/cm2, injections every 2 weeks, total number of injections: 3
  Other Names: Avastin
  Arms: HAART+ Bevacizumab injection

SUMMARY:
Kaposi sarcoma remains the most common malignancy among persons with HIV.

Lesions localized to the airway may cause bleeding, pain and dyspnea.

New therapeutic approaches for local disease are needed.

The purpose of this study is to compare the effectiveness of intralesional bevacizumab + HAART vs HAART alone in treating localized Kaposi´s sarcoma of the airway in patients with AIDS.

DETAILED DESCRIPTION:
Once disseminated disease is excluded, histologically confirmed HIV-positive patients with localized Kaposi's sarcoma of the airway will be randomized to receive HAART only or HAART + intralesional bevacizumab.

The primary outcome will be the size of lesions according to RECIST criteria. Patients in the HAART + bevacizumab arm will undergo series of 3 bevacizumab injections of 5 mg/cm3. Follow-up will be carried out through scheduled meetings for office setting examination every week for the first 8 weeks, then every 15 days for two months and finally every month for eight months.

Size of the lesions will be assessed by an independent observer and adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* KS of the oral cavity, pharynx and larynx, histopathologically confirmed
* HIV treatment-naïve

Exclusion Criteria:

* Airway obstructive lesions
* Actively bleeding lesions
* Tumor-associated oedema or ulceration
* Gastrointestinal KS
* KS in other nonnodal viscera

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Reyes-Teran, M.D., Study Director — Centro de Investigacion en Enfermedades Infecciosas; Yuria Ablanedo-Terrazas, M.D., Principal Investigator — Centro de Investigacion en Enfermedades Infecciosas
Locations (1):
- Centro de Investigacion en Enfermedades Infecciosas, México, State of Mexico, Mexico

REFERENCES:
- [Derived] Ablanedo-Terrazas Y, Alvarado-de la Barrera C, Ormsby CE, Ruiz-Cruz M, Reyes-Teran G. Intralesional bevacizumab in patients with human immunodeficiency virus-associated Kaposi's sarcoma in the upper airway. Laryngoscope. 2015 Apr;125(4):E132-7. doi: 10.1002/lary.24988. Epub 2014 Oct 27. PMID 25345840

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HAART | HAART+ Bevacizumab Injection
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HAART | HAART+ Bevacizumab Injection | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [24 to 32] | 35 [29 to 39] | 30.5 [24.7 to 38.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  Mexico | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Complete response will be assessed according to RECIST criteria
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- HAART; HAART+ Bevacizumab Injection: Bevacizumab: Intralesional bevacizumab, dosis of 5mg/cm2, injections every 2 weeks, total number of injections: 3
Arm/Group | HAART | HAART+ Bevacizumab Injection
Number analyzed (Participants) | 7 | 7
participants | 1 | 3

2. Secondary Outcome: Safety
Description: Adverse events will be assessed according to the Council for International Organizations of Medical Sciences (CIOMS) I Working Group the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Toxicity was graded and recorded using the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table)
Arm/Group | HAART | HAART+ Bevacizumab Injection
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAART (N=7) | HAART+ Bevacizumab Injection (N=7)
Fever (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — A patient had fever of 39°C after 3 days of receiving the first BVZ injection and starting ART. He was hospitalized and bronchoscopy revealed Mycobacterium avium complex pulmonary disease, so he was treated with clarithromycin and ethambutol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No